CLINICAL TRIAL: NCT02830230
Title: "Performance of HPV DNA Test in Presence of Co-infection With Common RTIs"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Sharmila Pimple, Dr Sharmila Pimple, Tata Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: 1671 RTIs And HPVDNA Test
Record Dates: First submitted 2016-06-29; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Cervical Inflammation and Human Papilloma Virus Performance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group/Case (Experimental): women with clinical cervicitis or cervicovaginitis as per NACO Guidelines will be enrolled in intervention group.
  women with clinical cervicitis or cervicovaginitis as per NACO Guidelines will be enrolled in intervention group.A cervico-vaginal swab shall be taken for Lab diagnosis of RTIs along with HPVDNA test on day 1.Women shall be treated with Tab Azithromycin 1gm and Tab Cefixime 400mg stat along with barrier contraception advised.The women will be followed up after 7-14 days .A repeat cervicovaginal swab and HPVDNA shall be repeated.
  Interventions: Drug: Tab cefixime,Tab Azithromycin
- Control group (No Intervention): Women without signs and symptoms of cervicitis or cervico-vaginitis.No intervention will be done in this group

INTERVENTIONS:
Drug: Tab cefixime,Tab Azithromycin — The women with clinical cervicitis will receive treatment for cervicitis.
  Arms: Intervention group/Case

SUMMARY:
There is a strong causal association between persisting genital tract infection with Human Papilloma Virus (HPV) and gradual progression of infection to cervical (mouth of uterus) cancer.The robust study from India have shown that single round of HPV DNA screening test to significantly reduce the cervical cancer mortality. The above findings are very encouraging since it demonstrates that a simple and reliable HPV DNA test which is now available in low income countries has a potential to be accepted as primary screening test in future.

The cross-sectional studies from developed countries from year 1999-2004 which focused to determine the test characteristics of HPV Hybrid Capture 2 test (HC2) to determine CIN2 and higher grade lesions, reported test sensitivity of 90% to 100% with a mean of 95%.

Similarly the cross-sectional studies from developing countries from 1993 to 2003 which have focused on test characteristics of HPV DNA Hybrid capture 2 (HC2) test to determine CIN2 and higher grade lesions has shown a sensitivity in the range of 50% to 91% with an average sensitivity of 79%.Among the developing countries cross-sectional study from India which evaluated test reported sensitivity of only 68.2%.

There is a statistical significant difference ( p value = 0.003) of sensitivity of HPV DNA HC2 test between the developed and developing countries to determine CIN2+ Lesions while there is no difference in the specificity.

A study that was conducted in Chinese women to detected the prevalence of HPV genotype among women with mucopurulent cervicitis, healthy women and women with Invasive cancer, the author reported a 10% higher failure rates to extract HPV DNA in cases of mucopurulent cervicitis as compared to other two groups.

So the study will explore if if the presence of untreated co-infections with STIs/RTIs (Sexually transmitted infections/Reproductive tract infections) resulting in cervical inflammation is somewhere interfering with low sensitivity of HC2 test due to presence of blood and excess mucus associated with the conditions leading to low sensitivity of the test in context to Indian Scenario.

DETAILED DESCRIPTION:
Methodology-The eligible women in the age group of 30-50 years will be screened. Eligibility criteria will be determined. Women with clinical cervicitis as per NACO guidelines on per speculum examination will been rolled as cases after signing the inform consent. Women with no signs and symptoms of cervicitis (No white discharge P/V,No lower Abdominal pain, No urinary symptoms,No dysperunia,No pruritis vulvae,No post coital bleeding)will be enrolled as controls after signing the inform consent. The participants ready to participate will be explained the details and the purpose of the study by Doctor.All the women enrolled in women shall be followed up after 7-14 days.

Day 1.Cervical swab from ectocervix and endocervix shall be collected. Additional vaginal swab Will be taken from lateral vaginal wall and posterior fornices for all women enrolled in study.The swabs will be evenly spread on a glass slide and heat fixed. The slides will be put in slide box to be transported to Microbiology Department for Gram staining for Gonococcal, Non-Gonococcal infections,Bacterial Vaginosis,Candida. Next, cervical cells for HPV DNA testing will be collected.

The women diagnosed with clinical cervicitis will receive treatment on the spot and advised use to use barrier contraception for 15 days.No treated will be given for the women in enrolled arm i.e women without clinical and lab STIs.

Day7-14- All the women enrolled in study shall be followed up after 7-14 days. Women will undergo per-speculum examination and clinical signs of cervicitis or cervicovaginitis will be reassessed again and documented.

A repeat cervical swab and vaginal swab shall be collected and send for gram staining for the above mentioned organisms.

A repeat, cervical cells for HPV DNA testing will be collected. Women who are positive for HPV DNA and STIs on follow up visits shall be counselled and referred for further evaluation and treatment to appropriate hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Sexually active women with clinically diagnosed cervicitis as per NACO guidelines will be enrolled as cases.
2. Sexually active women with no symptoms of STIs/RTIs and clinically no cervicitis will be enrolled as cases.

Exclusion Criteria:

1. Pregnant women.
2. Women not willing to follow up.
3. Not willing to use barrier contraception if diagnosed with STIs.
4. Women received antiboitics in last 4 weeks.
5. women with vaginitis without cervicitis on per speculum examination.
6. No drug allergy to the treating drugs.
7. No present or past history of cervical cancer. -

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 508 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Difference in the number of participants diagnosed with HPV infections before and after treating clinical cervicitis | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Reena J Wani, MD, Principal Investigator — HBT Medical College & R.N.Cooper Muncipal Hospital; Savita R Karnad, M.SC, Principal Investigator — HBT Medical College & R.N.Cooper Muncipal Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Tata Memorial Centre,Mumbai websiate — http://tmc.gov.in